CLINICAL TRIAL: NCT06394752
Title: UTERINE EVALUATION FOR THE IDENTIFICATION OF PATHOLOGY
Brief Title: UTERINE EVALUATION FOR THE IDENTIFICATION OF PATHOLOGY. This Study Will Compare the Intrauterine Pathology Detection Rate Between Standard of Care Hydrosonography, and a New Visual Saline Infusion Device Providing Direct Visualization of the Uterus.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Reproductive Health & Gynecology (Other)
Collaborators: Butterfly Biosciences, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TD-1033
Record Dates: First submitted 2024-04-25; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Hysteroscopy; Hysteroscopy Technique; Fertility Issues; Uterus Abnormal; Gynecology; Visualization; Infertility Female
Keywords: hysteroscopy; fertility; gynecology; hydrosonography; uterine evaluation; uterine pathology
MeSH Terms: conditions — Infertility; Uterine Anomalies; Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Visual Saline Infusion (Experimental): Visual Saline Infusion is intended to perform direct visual evaluation of the intrauterine space using a 2.7mm, steerable tip catheter with a camera.
  Interventions: Device: Visual Saline Infusion
- Hydrosonography (Active Comparator): Hydrosonography is the standard of care for intrauterine evaluation. It is performed by inserting a slim 2 mm catheter into the uterine cavity and infusing saline solution to expand the uterus, and using abdominal ultrasound to detect intrauterine pathology.
  Interventions: Device: Hydrosonography

INTERVENTIONS:
Device: Visual Saline Infusion — Visual Saline Infusion (VSI) is a new intrauterine imaging procedure to identify uterine pathology. The VSI device is a 2.7mm, steerable tip catheter with a camera and illumination at the distal end. The device is intended to evaluate the intrauterine space in an office based, outpatient setting using minimal volume of fluid (3-5cc's).
  Arms: Visual Saline Infusion
Device: Hydrosonography — Hydrosonography is an ultrasound based intrauterine imaging technique with sensitivity and specificity ranging from 90% to 100% for identifying uterine pathology. It is performed by inserting a slim 2 mm catheter into the uterine cavity and infusing saline solution to expand the uterus and using abdominal ultrasound to visualize the uterus.
  Arms: Hydrosonography

SUMMARY:
This is a prospective, single center, multiple arm cohort study intended to compare the diagnostic accuracy of a Visual Saline Infusion Device (VSI) device, vs standard of care Hydrosonography in reproductive aged women to identify pathology in the uterus.

DETAILED DESCRIPTION:
This is a prospective, single center, multiple arm cohort study intended to compare the diagnostic accuracy of a Visual Saline Infusion Device (VSI) device, vs standard of care Hydrosonography in reproductive aged women to identify pathology in the uterus.

Patients who are enrolled in the study will have a 1) Hydrosonography, and 2) Visual Saline Infusion procedure performed.

The Visual Saline Infusion Device is a 2.7mm, steerable tip catheter with a camera and illumination at the distal end. The device is intended to evaluate the intrauterine space in an office based, outpatient setting using minimal volume of fluid (3-5cc's).

This study will recruit up to 100 women from a fertility center in Los Angeles.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring a uterine cavity evaluation
2. Premenopausal women between ages of 18-45

Exclusion Criteria:

1. Positive test or history of any of the following conditions:

1a. Chlamydial pelvic infection

1b. Gonorrheal pelvic infection. 2. Positive Pregnancy Test 3. IUD currently in place

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Intrauterine pathology detection rate with Hydrosonography | Procedure of 2-5 minute duration
  The assessment will involve the examination of the intrauterine cavity for the presence of pathologies, including polyps, fibroids, adhesions, scar tissue, thickened endometrium, among others. The detection rate will be calculated as the ratio of the number of cases where abnormal pathologies are identified to the total number of cases examined.
Intrauterine pathology detection rate with Visual Saline Infusion | Procedure of approximately 2-5 minute duration
  The assessment will involve the examination of the intrauterine cavity for the presence of known pathologies, including polyps, fibroids, adhesions, scar tissue, thickened endometrium, among others. The detection rate will be calculated as the ratio of the number of cases where abnormal pathologies are identified to the total number of cases examined.

SECONDARY OUTCOMES:
Visual detection quality score (1-10) | Captured during procedure
  The visual detection quality score will be assessed using a normalized scale ranging from 1 (indicating poor or no visualization) to 10 (indicating excellent visualization), with scores assigned based on the clarity and detail of the intrauterine images obtained during the examination.
Fluid used during distention | Captured during procedure
  The volume of fluid used for distention of the uterus will be documented.
Pain during procedure | Collected on day of procedure
  The research team will interview the Subject and record the level of pain experienced based on the Wong Baker pain scale
Adverse events rate | Day of procedure and 24-48 hours post to procedure
  Anticipated and unanticipated adverse events will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Sam Najmabadi, MD, Principal Investigator — Center for Reproductive Health & Gynecology
Locations (2):
- Center for Reproductive Health & Gynecology, Beverly Hills, California, United States
- Punta Mita Fertility Center, Corral Del Risco, Nayarit, Mexico

IPD SHARING:
Plan to Share IPD: Undecided